CLINICAL TRIAL: NCT03701594
Title: The Impact of Yoga-based Physical Therapy on Heart Rate Variability for Individuals With Traumatic Brain Injury: a Pilot Study
Brief Title: The Impact of Yoga-based Physical Therapy for Individuals With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, David Ripley, Medical Director, Brain Injury Medicine and Rehabilitation, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Yoga and HRV
Record Dates: First submitted 2018-10-04; First posted 2018-10-10 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, controlled, single-blinded, crossover design with three conditions: condition A will consist of 1 hour of yoga-based physical therapy session in a group setting; condition B will consist of 1 hour of one-on-one conventional physical therapy; condition C will consist of 1 hour of seated rest in a relaxing environment in a group setting.
Who Masked: Outcomes Assessor
Masking Description: The people administering the self-reported outcome measures will be blinded to the condition the subject participated in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga-based physical therapy group (Experimental): The yoga-based physical therapy session will take place in an enclosed, quiet space to minimize outside noise or distraction. The lights will be dimmed, and light, instrumental, calming music will be played throughout. The group will consist of approximately 2-5 individuals depending on the physical capabilities and assistance levels required. The session will consist of an introduction to pranayama (foundational breath-based exercises) followed by asanas, or physical postures, that will be modified according to each individual's physical abilities. The session will close with a 4-5 minute savasana performed in a supine or seated position pending patient physical abilities, which consists of progressive relaxation, guided meditation, and guided motor imagery.
  Interventions: Other: Yoga-based physical therapy group
- Seated rest (Active Comparator): Subjects will engage in 1 hour of seated rest in a relaxing environment in a group of approximately 2-5 individuals. This session will occur in the same enclosed, quiet space as condition A to minimize outside noise or distraction and to reproduce environment of condition A. The lights will be dimmed, and the same light, instrumental, calming music will be played throughout to contribute to a relaxing ambiance. Subjects will be instructed to rest quietly.
  Interventions: Other: Seated Rest
- Conventional Physical Therapy (Active Comparator): Subjects will engage in 1 hour of a conventional PT session (or "treatment as usual") led by a different physical therapist than who is leading the yoga-based session to minimize bias. There will be no restrictions on what can and cannot occur during conventional PT sessions in order to accurately represent and preserve the wide range of treatments that may occur during a physical therapy session in the inpatient setting. Examples of what may occur include, but are not limited to: gait, standing balance, functional mobility, or therapeutic exercise.
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Yoga-based physical therapy group — All yoga-based sessions will be led by the same therapist to maximize between-session consistency. A trained researcher will also be present to provide additional cueing to subjects when required. The basic elements of the postures are similar to that of traditional physical therapy balance exercises. Cues will be provided throughout to pair appropriate breath cycles with appropriate postures consistent with a standard, able-bodied yoga program. The session will close with a 4-5 minute savasana performed in a supine or seated position pending patient physical abilities, which consists of progressive relaxation, guided meditation, and guided motor imagery.
  Arms: Yoga-based physical therapy group
Other: Seated Rest — Subjects will engage in 1 hour of seated rest in a relaxing environment in a group of approximately 2-5 individuals. This session will occur in the same enclosed, quiet space as condition A to minimize outside noise or distraction and to reproduce environment of condition A. The lights will be dimmed, and the same light, instrumental, calming music will be played throughout to contribute to a relaxing ambiance. Subjects will be instructed to rest quietly.
  Arms: Seated rest
Other: Conventional Physical Therapy — Subjects will engage in 1 hour of a conventional PT session (or "treatment as usual") led by a different physical therapist than who is leading the yoga-based session to minimize bias. There will be no restrictions on what can and cannot occur during conventional PT sessions in order to accurately represent and preserve the wide range of treatments that may occur during a physical therapy session in the inpatient setting. Examples of what may occur include, but are not limited to: gait, standing balance, functional mobility, or therapeutic exercise.
  Arms: Conventional Physical Therapy

SUMMARY:
This study aims to explore if a yoga-based physical therapy session would promote improved (increased) heart rate variability in subjects with traumatic brain injuries. The results of this pilot study may inform a larger-scale study of the effects of regular participation in a yoga-based program as an adjunct to traditional physical therapy. The secondary objective is to determine whether a yoga-based physical therapy session would impact anxiety, fatigue, or agitation and/or sleep quality. The study will enroll up to 30 inpatient subjects on a rolling basis as they are admitted with traumatic brain injury over a 12 month period at the Shirley Ryan AbilityLab.

Each person in the study will participate in three conditions in a random order across three days: 1 hour of yoga-based physical therapy session in a group setting,1 hour of one-on-one conventional physical therapy, and 1 hour of seated rest in a relaxing environment in a group setting.

The hypothesis is that individuals who participate in 1 hour of a yoga-based physical therapy session in a group setting will demonstrate a significant improvement in heart rate variability, anxiety, fatigue, and agitation after the session when compared to the same measures after 1 hour of a conventional physical therapy session and 1 hour of seated rest in a relaxing environment. Sleep will also be assessed with an activity monitor.

DETAILED DESCRIPTION:
Admissions to the traumatic brain injury service of Shirley Ryan AbilityLab will be reviewed on a weekly basis, and eligible patients will be approached to attain assent/consent. Patients will be randomized as to which condition they participate in first. Subjects will be instructed not to eat or drink caffeine within 1 hour of participating in a condition. A trained researcher will apply three sensors to the chest. The sensors to monitor heart rate variability (HRV) via electrocardiogram (EKG) are from the BioStampRC Discovery Kit MC10, Inc., and are research-grade, non-invasive, wireless, wearable sensors. For each sensor location, the skin will be prepped and cleaned using alcohol wipes. Sensors are placed on the skin using adhesive stickers that minimize irritation. Medical dressing (Tegaderm, 3M) may also be used to ensure adhesion and proper contact with the skin. Sensors will be cleaned with soap and water before and after use. Vital signs will be measured. The self-reported outcome measures will be administered by a blinded clinician.

The subject will participate in the assigned condition for that day as determined by randomization, and HRV will be monitored throughout the condition. Immediately following the 1-hour condition, the sensors will be removed by a trained researcher and the self-reported outcomes will again be administered under the supervision of a blinded clinician. Subjects will complete forms as able, but if they require physical assistance to fill out or verbal assistance in reading the questions, such assistance will be provided. Sleep quality will be captured by an activity monitor. Research staff will don and doff the activity monitors.

All sessions will be supervised by a physical therapist. Research staff will be responsible for all sensor recording practices, such as instrumenting the sensors and marking therapy activities on a computer tablet using the BioStampRC software. Research staff will also keep a written log of activities as they are undertaken during the assessments, including notable events, amount and type of assistance, or use of external devices. Logs will be consulted during analysis to compare with the timestamped sensor data.

Audio/video recording may be utilized in order to allow a registered yoga therapist to validate the yoga-based program led by the researcher-clinician physical therapist. The recordings would only be viewed by the physical therapist and registered yoga therapist, and destroyed after publication of the research. The videos would be stored in a password-protected device; the yoga therapist and physical therapist would be the only individuals with access.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with traumatic brain injury admitted to the Shirley Ryan AbilityLab (SRALab)
* Age 18 or older
* Able and willing to give written consent or has an identified medical proxy willing to give written consent on behalf of the individual
* Able to follow commands consistently with a reasonable amount of verbal or visual cues in order to participate in a 60-minute physical therapy session in a group setting
* Able to attend to a task with reasonable amount of verbal or visual cues in order to participate in a 60-minute physical therapy session in a group setting
* Behaviorally appropriate for a group setting in terms of verbal or physical escalation/aggression

Exclusion Criteria:

* Serious cardiac conditions (arrhythmias) or neurological comorbidities (such as multiple sclerosis, Alzheimer's disease, Parkinson's disease, etc.)
* Pregnant or nursing
* Skin allergies or irritation; open wounds in the areas that the sensors would be applied to
* Utilizing a powered, implanted cardiac device for monitoring or supporting heart function (i.e. pacemaker, defibrillator, or LVAD)
* Non-English speaking patients, due to necessity for an interpreter to be present constantly interpreting, which could impact the low-stimulation setting of the intervention
* Aphasia or any difficulties in accurately self-reporting

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | The sensors will be worn throughout the three 1 hour long conditions.
  Heart rate variability will be measured by MC-10 sensors placed on the chest.

SECONDARY OUTCOMES:
State-Trait Anxiety - 6 Question Version | This measure will be administered before and after each condition (yoga, conventional PT, seated rest). Data will be analyzed within approximately 10 months from enrollment of first participant, and research publication will be pursued.
  Score range: 6-24. This measure allows for assessment of self-reported present-state anxiety. It is a 6-question version of a longer original questionnaire that will aide in preventing cognitive fatigue that can sometimes be faced with longer surveys.
Global Fatigue Index-Modified | This measure will be administered before and after each condition (yoga, conventional PT, seated rest). Data will be analyzed within approximately 10 months from enrollment of first participant, and research publication will be pursued.
  Score range: 3-15. A shortened version of the original global fatigue index with modified language to reflect present-state feelings will be utilized to measure present-state fatigue.
Agitated Behavior Scale | This measure will be administered before and after each condition (yoga, conventional PT, seated rest) only if the person presents with agitation. Data will be analyzed within approximately 10 months from enrollment of first participant.
  Score range: 14-56 (higher=more agitated). This outcome will only be collected when the patient presents with agitation and is actively being assessed with the Agitated Behavior Scale (ABS) on a regular basis by the nursing staff. The ABS measures behavioral aspects of agitation during the acute phase of recovery from acquired brain injury including aspects of aggression, disinhibition, and lability.

CONTACTS AND LOCATIONS:
Overall Officials: David Ripley, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Krese K, Ingraham B, O'Brien MK, Mummidisetty CK, McNulty M, Srdanovic N, Kocherginsky M, Ripley D. The impact of a yoga-based physical therapy group for individuals with traumatic brain injury: results from a pilot study. Brain Inj. 2020 Jul 2;34(8):1118-1126. doi: 10.1080/02699052.2020.1776394. Epub 2020 Jun 12. PMID 32530717